CLINICAL TRIAL: NCT00893867
Title: A Double Blind, Randomized, Placebo-controlled, Parallel Group, Multicenter Phase 3 Pivotal Study to Assess the Safety and Efficacy of 1mg/kg/Day Intravenous DP-b99 Over 4 Consecutive Days Versus Placebo When Initiated Within Nine Hours of Acute Ischemic Stroke Onset
Brief Title: Efficacy and Safety Study of DP-b99 in Treating Acute Ischemic Stroke
Acronym: MACSI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The result of a pre-planned interim futility analysis
Sponsor: D-Pharm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ptcl-01373
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; neuroprotective agent
MeSH Terms: conditions — Ischemic Stroke | interventions — DP-b99

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DP-b99 (Experimental)
  Interventions: Drug: DP-b99
- Mannitol (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DP-b99 — 1mg/kg/day over 4 consecutive days given intravenously and initiated up to 9 hours following acute stroke onset.
  Arms: DP-b99
Drug: Placebo — 1mg/kg/day over 4 consecutive days given intravenously and initiated up to 9 hours following acute stroke onset.
  Arms: Mannitol

SUMMARY:
The purpose of this trial is to determine if intravenous administration of the metal ion trapping agent DP-b99 up to 9 hours following acute ischemic stroke onset, and then for 3 additional days (4 consecutive days in total) is effective in improving long term outcome. Patients will be followed up for 3 months after the stroke.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled, multicenter, multi-national, parallel-arm, pivotal study comparing a placebo group to a DP-b99 group treated with intravenous 1.0 mg/kg/d for 4 consecutive days, in acute ischemic stroke patients with an entry National Institutes of Health Stroke Scale (NIHSS) score of 10-16 and a clinical syndrome that includes at least 1 of the following: language dysfunction, visual field defect or Extinction and Inattention (formerly Neglect) (as reflected by at least 1 point on any of the corresponding items of the NIHSS: 9, 3 or 11). An interim analysis for futility will be performed after Day 90 (or last available observation) primary endpoint data have been collected on about 45% of subjects planned to be enrolled. Clinical trial material (CTM) will be administered within 9 hours after the onset of acute ischemic stroke symptoms. Subjects will be randomized at a ratio of 1:1 to receive either DP-b99 or placebo. A data and safety monitoring board (DSMB) will assess the accumulating safety data periodically and will oversee the interim futility analysis.

ELIGIBILITY:
Inclusion criteria:

1. M or F age 18 - 85, inclusive
2. Suffered an acute, likely hemispheric, ischemic stroke, defined as acute, focal, neurological deficit(s), secondary to a presumed vascular event, which must include at least one of the following components (as reflected by at least 1 point on any of the corresponding items of the NIHSS: 3, 9 or 11):

   * Visual
   * Best Language
   * Extinction and Inattention (formerly Neglect)
3. Suffered the onset of an acute ischemic stroke that can be evaluated and treatment initiated within 9 hours after the onset of acute ischemic stroke symptoms.
4. Screening NIHSS score of 10 to 16, inclusive
5. Readily accessible peripheral venous access for clinical trial material (CTM) administration and blood sampling
6. Ability to understand the requirements of the study and be willing to provide written informed consent as evidenced by signature on an informed consent document approved by an institutional review board or independent ethics committee, and agree to abide by the study restrictions and return for the required assessments.
7. Provided written authorization for use and disclosure of protected health information in accordance with the Health Insurance Portability and Accountability Act in the United States and the Personal Information Protection and Electronic Documents Act in Canada

Exclusion Criteria:

1. An intracerebral or subarachnoid hemorrhage per screening/baseline computerized tomography scan or susceptibility-weighted magnetic resonance imaging
2. A candidate for either:

   1. thrombolytic therapy, or have been treated with thrombolytic therapy for the current stroke
   2. mechanical thromboembolectomy, or have been treated with mechanical thromboembolectomy for the current stroke
3. Delirious, comatose or stuporous or demented, or having a mental impairment that in the investigator's opinion renders the subject incapable to participate in the study
4. Have seizure(s) anytime from stroke onset to screening/baseline NIHSS evaluation
5. Neurological or non-neurological comorbidities that in the investigator's opinion may lead, independent of the current stroke, to further deterioration in the subject's neurological status during the trial period, or may render the study's neurological assessments inconclusive for the purpose of evaluating solely the stroke's effects
6. Likely to undergo a procedure involving cardiopulmonary bypass during the study period
7. Suffered a myocardial infarction in the last 90 days
8. Any medical condition that in the investigator's opinion may threaten the subject's ability to complete the study (e.g., concurrent significant or life-threatening diseases, such as malignancies or end stage organ failure)
9. Rapid spontaneous improvement of neurological signs during screening/baseline assessments
10. Premorbid neurological deficits and functional limitations assessed by a pre-stroke Modified Rankin Scale score of > 1
11. Suffered a stroke within 90 days of the screening/baseline assessments that is either diagnostically confirmed or assumed to be in the same cerebral territory as is the current acute stroke
12. Either severe hypertension or hypotension, as measured by at least 2 consecutive supine measurements taken 10 minutes apart prior to randomization.
13. Significant current renal or hepatic disease(s): a serum creatinine concentration of >2.5 mg/dL; alanine aminotransferase, aspartate aminotransferase, or gamma-glutamyl transferase values that are three times greater than the upper limit of normal.
14. Have a platelet count of <100,000/mm3 or, for patients on oral anticoagulants at study entry, INR of >4
15. Female of childbearing potential who is not willing to use adequate and effective birth control measures for the duration of the trial. Effective birth control measures include hormonal contraception, a barrier method such as a diaphragm, intrauterine device and/or condom with spermicide
16. Positive urine pregnancy test at screening/baseline or be a lactating female
17. Currently dependent on, or abusing, alcohol or one or more of the following: sympathomimetic amines, cannabis, cocaine, hallucinogens, inhalants, opioids, phencyclidine, sedatives and hypnotics
18. Received an investigational drug or product or participated in an investigational drug study within a period of 30 days prior to receiving study medication or have previously participated in a clinical trial involving DP-b99
19. Severe anemia as measured by a hemoglobin value of < 7 g/dl.
20. In a dependent relationship with the physician or the study sponsor.
21. Known hypersensitivity to any component of the investigational product.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2009-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) categorical analysis ("shift") | 90 days

SECONDARY OUTCOMES:
Recovery, defined as a score of ≤ 1 on modified Rankin Score | 90 days
Safety and tolerability | throughout study - baseline until day 90
  the numbers of patients with treatment-emergent adverse events, results of physical examination, 12-lead electrocardiogram, vital signs and laboratory tests (complete blood count, chemistry and urinalysis)
recovery as assessed by an NIHSS of not more than 1 | 90 days
'home time' | 90 days
  exploratory endpoint of 'home time', which measures the length of time (as number of nights)spent at home/relatives' home between hospital discharge and day 90

CONTACTS AND LOCATIONS:
Overall Officials: Ashfaq Shuaib, MD, Principal Investigator — University of Alberta Hospital, Edmonton, Canada; Vasco Salgado, MD, Principal Investigator — Hospital Professor Doutor Fernando Fonseca, EPE, Amadora, Portugal; Philippe Lyrer, Prof. Dr., Principal Investigator — Universitätsspital Basel, Neurologie, Basel, Switzerland; Tobien Schreuder, MD, Principal Investigator — Atrium MC Parkstad, Heerlen, Netherlands; Maria S Rocha, MD, Principal Investigator — Hospital Santa Marcelina, Sao Paulo, Brasil; Hugues Chabriat, Prof., Principal Investigator — Hôpital Lariboisière - Service Neurologie, Paris, France
Locations (154):
- United States (13):
  - Research Center of Southern California, Oceanside, California
  - Associated Neurologists, P.C., Danbury, Connecticut
  - Memorial Health University Medical Center, Savannah, Georgia
  - The University of Kentucky The Methodist Hospital, Lexington, Kentucky
  - University of Louisville, Kentucky Neuroscience Research, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Capital Health Regional Medical Center Neuroscience Institute, Trenton, New Jersey
  - Presbitarian Hospital, Charlotte, North Carolina
  - St. Elizabeth's Medical Center, Youngstown, Ohio
  - Legacy Meridian Park Medical Center, Tualatin, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The Methodist Hospital, Houston, Texas
  - Carilion Clinic, Roanoke, Virginia
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck
  - Landeskrankenhaus Klagenfurt, Klagenfurt
  - Abt. Neurologie und Psychiatrie, Linz
  - LKH St. Pölten Department of Neurology, Sankt Pölten
- Brazil (9):
  - Santa Casa de Misericordia de Belo Horizonte Departamento de Neurologia, Belo Horizonte
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Hospital Moinhos de Vento, Porto Alegre
  - Hospital Mãe de Deus, Porto Alegre
  - Santa Casa de Misericórdia de Porto Alegre Policlinica Santa Clara Sala de Neurologia, Porto Alegre
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto Unidade de Emergência Centro de Estudos, Ribeirão Preto
  - Hospital São José de Joinville, Santa Catarina
  - Hospital Santa Marcelina, São Paulo
  - UNIFESP, São Paulo
- Canada (7):
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Grey Nun's Community Hospital, Edmonton
  - University of Alberta Hospital, Edmonton
  - Hamilton Health Sciences Centre, Hamilton
  - Kingston General Hospital, Kingston
  - Chinook Regional Hospital, Lethbridge
  - CHA- Hôpital de l'Enfant-Jésus, Québec
- Czechia (8):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Clinic of Neurology, Hradec Králové
  - Hospital Jihlava Clinic of Neurology, Jihlava
  - Hospital Vítkovice Clinic of Neurology, Ostrava
  - County Hospital Pardubice Clinic of Neurology, Pardubice
  - Clinic of Neurology, Stroke Center, Charles University, Prague
  - University Hospital Kralovske Vinohrady, Prague
  - University Hospital Motol Clinic of Neurology, Prague
- France (7):
  - CHU Jean Minjoz Besançon, Besançon
  - Hopital Pellegrin-Tripode, Bordeaux
  - CHU Henri Mondor, Créteil
  - Hopital Gui de Chauliac, Montpellier
  - Hôpital Bichat, Paris
  - Hôpital Lariboisière - Service Neurologie, Paris
  - Hôpital Saint Jean, Perpignan
- Germany (27):
  - Ärztlicher Direktor Neurologische Klinik, Neurologische Klink GmbH der Rhoen-Klinikum AG, Bad Neustadt / Saale
  - Marien-Krankenhaus gGmbH, Abteilung für Neurologie, Bergisch Gladbach
  - DRK Kliniken Berlin, Klinik fuer Neurologie, Berlin
  - Vivantes Klinikum Neukölln, Klinik für Neurologie, Stroke Unit, Berlin
  - Klinikum Bremen-Mitte, Bremen
  - Klinikum Bremerhaven-Reinkenheide gGmbH, Neurologische Klinik, Bremerhaven
  - Klinikum Chemnitz GmbH Chefarzt Klinik für Neurologie, Chemnitz
  - Klinikum Köln Merheim, Department of Neurology, Cologne
  - Helios Klinikum Erfurt GmbH, Erfurt
  - Universitätsklinikum Erlangen, Neurologische klinik, Erlangen
  - Universitätsklinikum Essen, Klinik und Poliklinik für Neurologie, Essen
  - Neurologische Universitätsklinik Freiburg, Neurozentrum, Freiburg im Breisgau
  - Klinikum Fulda, Neurologische Klinik, Fulda
  - Evangelische Kliniken Gelsenkirchen GmbH Klinik für Neurologie und Klinische Neurophysiologie, Gelsenkirchen
  - Georg-August-Universitat Gottingen Neurologische Klinik, Göttingen
  - Ernst Moritz Arndt University, Grifswald
  - Askepios Klinik Altona, Hamburg
  - Askepios Klinik Heidberg, Hamburg
  - Universitätsklinikum Leipzig AöR, Klinik und Poliklinik für Neurologie, Leipzig
  - Klinikum der Otto-von-Guericke-Universität Magdeburg, Neurologische Universitätsklinik, Magdeburg
  - Johannes Gutenberg Universitat, Klinik und Poliklinik fur Neurologie, Mainz
  - Klinikum 1 Minden, Neurologische Klinik, Minden
  - Universität Rostock Chefarzt Abteilung Neurologie, Rostock
  - ASKLEPIOS Fachklinikum Teupitz, Teupitz
  - Krankenhaus der Bramherzigen Brüder, Trier
  - Universitätsklinikum Ulm, Abteilung für Neurologie im RKU, Ulm
  - Heinrich Braun Klinikum Zwickau, Zwickau
- Hungary (9):
  - Fővárosi Önkormányzat Péterfy Sándor utcai Kórház- Rendelőintézet és Baleseti Központ, Budapest
  - Állami Egészségügyi Központ, Budapest
  - Kenezy Korhaz Rendelointezet Egezsegugyi Szolgaltato Nonprofit Kft., Debrecen
  - University of Debrecen, Medical and Health Science Center, Debrecen
  - Aladár Petz County Teaching Hospital, Győr
  - PM Flór Ferenc County Hospital, Kistarcsa
  - Borsod-Abaúj-Zemplén County Hospital Miskolc, Miskolc
  - Pécsi Tudományegyetem Klinikai Központ, Pécs
  - Zala Megyei Kórház, Zalaegerszeg
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - Neurological Dept. Edith Wolfson Medical Center, Holon
  - Meir Medical Center, Kfar Saba
  - Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (12):
  - Ospedale Regionale Valle d'Aosta, Aosta
  - Dipartimento di Neuroscienze, Ospedale di Brotzu, Cagliari
  - Ospedale di Circolo di Varese, Lombardia
  - Istituto Scientifico San Raffaele - Stroke Unit, Milan
  - Istituto Neurologico C. Mondino, Pavia
  - Università di Perugia, Division of Internal and Cardiovascular Medicine - Stroke Unit, Perugia
  - Presidio Ospedaliero di Piacenza, Piacenza
  - Azienda Ospedaliera Sant'Andrea, Stroke Unit, Rome
  - Istituto Patologia Generale U.C.S.C, Rome
  - U.O.C. Stroke Unit, Rome
  - Università di Roma "La Sapienza" - Stroke Unit, Rome
  - Azienda Ospedaliera Universitaria "Santa Maria della Misericordia" Stroke Unit, Udine
- Netherlands (4):
  - Catharina Ziekenhuis Neurologie, Eindhoven
  - Medisch Spectrum Twente Hoofd Afdeling Vasculaire Neurologie, Enschede
  - Atrium MC Parkstad, Heerlen
  - Isala Klinieken Ploikliniek Neurologie, Zwolle
- Poland (9):
  - Pomerania Traumatology Center, Regional Specialist Hospital im. Nicolaus Copernicus, Gdansk
  - Medical University of Lublin, Department of Neurology, Stroke Unit, Lublin
  - Samodzielny Publiczny Zespol Zakladow Opieki Zdrowotnej w Sandomierzu, Sandomierz
  - Szpital Powiatowy im. Marii Curie - Skłodowskiej w Skarżysku-Kamiennej, Skarżysko-Kamienna
  - Wojewodzki Szpital Specjalistyczny Nr 1 im. Prof. Jozefa Gasinskiego, Tychy
  - Instytut Psychiatrii i Neurologii Oddział Neurologiczny z Pododdziałem Udarowym, Warsaw
  - Medical University of Warsaw, Department of Neurology, Warsaw
  - Szpital Wolski im. dr Anny Gostyńskiej Samodzielny Publiczny Zakład Opieki Zdrowotnej, Oddział Neurologii, Warsaw
  - Wojskowy Instytut Medyczny, Oddział Neurologii, Warsaw
- Portugal (5):
  - Hospital Professor Doutor Fernando Fonseca, EPE, Amadora
  - Centro Hospitalar de Coimbra EPE, Coimbra
  - Hospitais da Universidadde de Coimbra, EPE, Coimbra
  - Centro de Estudos Egas Moniz - Hospital de Santa Maria, Lisbon
  - Hospital de São Sebastião, EPE, Santa Maria da Feira
- Slovakia (5):
  - Neurology Clinic, Faculty Hospital in Martin, Martin
  - University Hospital Nitra, Nitra
  - Hospital un Poliklinic, Spišská Nová Ves
  - Faculty Hospital Trnava, Trnava
  - Neurology dept.,Hospital Zilina, Žilina
- South Africa (6):
  - Fichmed, Bloemfontein
  - Constantiaberg Medi-clinic, Cape Town
  - Union Hospital, Gauteng
  - Helderberg Research Institute, Western Cape
  - Triervlei Trial Centre, Western Cape
  - Clinical Projects Research, Worcester
- South Korea (9):
  - Dong-A Medical Center, Busan
  - Inje University BUSAN Paik Hospital, Busan
  - Inje University ILSAN Paik Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - ASAN Medical Center, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's hospital, Seoul
- Spain (13):
  - Hospital Universitario de Albacete, Albacete
  - Hospital De La Santa Ta Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Germans Triasy Pujol, Barcelona
  - Hospital Vall D'hebron, Barcelona
  - Hospital Gregorio Maranon, Madrid
  - Hospital La Princesa, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Consorcio Hospital General Universitario Valencia, Valencia
  - Hospital Clinico Universitario De Valladolid, Valladolid
- Switzerland (2):
  - Universitätsspital Basel, Neurologie, Basel
  - Universitätsspital Zürich, Klinik für Neurologie, Zurich

REFERENCES:
- [Background] Diener HC, Schneider D, Lampl Y, Bornstein NM, Kozak A, Rosenberg G. DP-b99, a membrane-activated metal ion chelator, as neuroprotective therapy in ischemic stroke. Stroke. 2008 Jun;39(6):1774-8. doi: 10.1161/STROKEAHA.107.506378. Epub 2008 Apr 10. PMID 18403736
- [Background] Rosenberg G, Angel I, Kozak A. Clinical pharmacology of DP-b99 in healthy volunteers: first administration to humans. Br J Clin Pharmacol. 2005 Jul;60(1):7-16. doi: 10.1111/j.1365-2125.2005.02378.x. PMID 15963088
- [Background] Barkalifa R, Hershfinkel M, Friedman JE, Kozak A, Sekler I. The lipophilic zinc chelator DP-b99 prevents zinc induced neuronal death. Eur J Pharmacol. 2009 Sep 15;618(1-3):15-21. doi: 10.1016/j.ejphar.2009.07.019. Epub 2009 Jul 19. PMID 19622352
- [Background] Rosenberg G, Bornstein N, Diener HC, Gorelick PB, Shuaib A, Lees K; MACSI investigators. The Membrane-Activated Chelator Stroke Intervention (MACSI) Trial of DP-b99 in acute ischemic stroke: a randomized, double-blind, placebo-controlled, multinational pivotal phase III study. Int J Stroke. 2011 Aug;6(4):362-7. doi: 10.1111/j.1747-4949.2011.00608.x. Epub 2011 Jun 6. PMID 21645269
- [Background] Rosenberg G, Marshall LS, Caraco Y. The neuroprotective agent DP-b99 does not interact with s-warfarin in vivo despite significant CYP2C9 inhibition in vitro. Basic Clin Pharmacol Toxicol. 2011 Apr;108(4):289-92. doi: 10.1111/j.1742-7843.2010.00654.x. Epub 2010 Dec 16. No abstract available. PMID 21414144